CLINICAL TRIAL: NCT01167010
Title: A Phase III, Randomized, Non-inferiority, Open-label, Comparative Study Between Foraseq® Inhalation Capsules, Eurofarma's Single Formoterol / Budesonide Inhalation Capsule and Single Alenia® Inhalation Capsule in Asthmatic Patients
Brief Title: A Non-inferiority, Comparative Study Between Foraseq®, Eurofarma´s Formoterol/Budesonide and Alenia® in Asthma
Acronym: UNIK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF111
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Formoterol/Budesonide (Experimental): formoterol and budesonide will be administered at the 12/400 µg dosage, twice a day for 12 weeks.
  Interventions: Drug: Formoterol/Budesonide
- Foraseq (Active Comparator): Foraseq will be administered at the 12/400 µg dosage, twice a da for 12 weeks.
  Interventions: Drug: Foraseq
- Alenia (Active Comparator): Alenia will be administered at the 12/400 µg dosage, twice a da for 12 weeks.
  Interventions: Drug: Alenia

INTERVENTIONS:
Drug: Formoterol/Budesonide — formoterol and budesonide will be administered at the 12/400 µg dosage, twice a da for 12 weeks.
  Arms: Formoterol/Budesonide
Drug: Foraseq — foraseq will be administered at the 12/400 µg dosage, twice a da for 12 weeks.
  Other Names: Formoterol/Budesonide
  Arms: Foraseq
Drug: Alenia — Alenia will be administered at the 12/400 µg dosage, twice a da for 12 weeks.
  Other Names: Formoterol/Budesonide
  Arms: Alenia

SUMMARY:
The primary objective will be to compare the Eurofarma and Alenia formulations regarding their impact on the pulmonary function of mild to moderate persistent asthma patients and the secondary objective will be to compare the three study formulations regarding the clinical control of the symptoms and the patients' compliance to the treatment.

DETAILED DESCRIPTION:
The primary objective will be to compare the Eurofarma and Alenia formulations regarding their impact on the pulmonary function of mild to moderate persistent asthma patients and the secondary objective will be to compare the three study formulations regarding the clinical control of the symptoms and the patients' compliance to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign the ICF;
* ≥ 12 years old;
* Have a diagnosis of mild to moderate persistent asthma diagnosis, as per the GINA classification (www.ginasthma.com),18 with symptoms for at least 6 months and clinically stable for at least 1 month with the ACQ-7 test <3,0;
* Current use of inhaled corticosteroid (equivalent to 1000 µg of beclomethasone dipropionate) whether associated or not with long-term β2 adrenergics and relief medication (salbutamol or equivalent);
* Initial FEV1 of at least 50% of the normal value expected;
* Serum cortisol evaluation within the normal limits

Exclusion Criteria:

* Use of oral or parenteral corticosteroid within the last 3 months before the study;
* Hospitalization needed due to asthma within the last 3 months before the study;
* Active smokers, defined as the consumption of cigarettes, pipes, cigars, or any other form of smoking in any amount within the last 3 months;
* Presence of serious co-morbidities, such as cardiovascular, renal, liver, neurological, neoplastic, hematological, infectious, dermatologic, neurological, or psychiatric disease, or chronic respiratory disease other than asthma;
* Recent participation (<6 months) or expected participation in other clinical trials involving drug products of any nature or in studies consisting of any form of intervention for the treatment of asthma;
* Intolerance or allergy to any component of the drugs evaluated in the study;
* Pregnant or lactating women;
* Chronic use of routine β-blockers orally or intravenously, including ophthalmic solutions.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Centro de Referencia em Enfermidades Respiratoria e Alergica, Salvador, Estado de Bahia
  - Hospital de Clinicas UFPR, Curitiba, Paraná
  - IMA Brasil - Instituto de Pesquisa Clínica e Medicina Avançada, São Paulo, São Paulo
  - Stelmach Pesquisa Clinica, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila, Sorocaba, São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Foraseq: Foraseq will be administered at the 12/400 µg dosage, twice a day for 12 weeks.
- Alenia: Alenia will be administered at the 12/400 µg dosage, twice a day for 12 weeks.
Period: Overall Study
Arm/Group | Formoterol/Budesonide | Foraseq | Alenia
Started | 184 | 184 | 184
Completed | 154 | 145 | 151
Not Completed | 30 | 39 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol/Budesonide | Foraseq | Alenia | Total
Number analyzed (Participants) | 154 | 145 | 151 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 25 | 21 | 74
  Between 18 and 65 years | 119 | 112 | 121 | 352
  >=65 years | 7 | 8 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (17) | 39 (17) | 39 (16) | 39 (17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The protocol population (PP) consisted of all patients who adhered to the study procedures and treatment did not violate selection criteria, did not presented other major protocol violations according to the criteria of who had FEV1 data at the final study visit (primary endpoint effectiveness).
  Participants
    Female | 99 | 99 | 110 | 308
    Male | 55 | 46 | 41 | 142
Region of Enrollment [Number; unit: participants]
  Brazil | 154 | 145 | 151 | 450

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at the Final Visit (FV)
Description: The primary efficacy analysis was performed by evaluating non-inferiority of Eurofarma's device compared to Alenia® in relation to FEV1 (in liters) in FV in the PP population
Time Frame: 12 weeks
Population: The study aims to demonstrate the non-inferiority of the FEV1 (in liters) at the final visit (FV) in the per-protocol (PP) population results for the Formoterol/Budesonide product compared to Alenia.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Formoterol/Budesonide | Alenia
Number analyzed (Participants) | 154 | 150
Liter | 2.53 (0.79) | 2.51 (0.77)

2. Secondary Outcome: FEV1 (L) in VF in the ITT Population, to Assess the Difference Between the Three Groups
Description: The mean FEV1 (L) in VF were compared between the three groups using the nonparametric Kruskal-Walllis test and the ITT population. A nonparametric test was used since the variable did not show normal distribution in the Foraseq® group.
Time Frame: 12 weeks
Population: FEV1 (L) measurement at the final study visit (FV) considering the comparison of non-inferiority of Eurofarma research product with Foraseq®, FEV1 (L) of the ITT population.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Alenia | Formoterol/Budesonide | Foraseq
Number analyzed (Participants) | 150 | 154 | 145
Liter | 2.49 (0.77) | 2.52 (0.80) | 2.46 (0.88)

ADVERSE EVENTS:
Arm/Group | Formoterol/Budesonide | Foraseq | Alenia
Serious Adverse Events (participants affected / at risk) | 1/154 | 0/145 | 0/151
Other Adverse Events (participants affected / at risk) | 1/154 | 0/145 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formoterol/Budesonide (N=154) | Foraseq (N=145) | Alenia (N=151)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Thrombocytopenia
Leukopenia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Leukopenia
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Formoterol/Budesonide (N=154) | Foraseq (N=145) | Alenia (N=151)
Left and posterior knee trauma infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other